CLINICAL TRIAL: NCT06747728
Title: Bevacizumab Neoadjuvant Therapy for New High-grade Gliomas in the Brain
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The First Affiliated Hospital of Zhengzhou University (Other)
Responsible Party: Principal Investigator, Junkuan Wang, Clinical Professor, The First Affiliated Hospital of Zhengzhou University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: QLMA-GBM-IIT-101
Record Dates: First submitted 2024-12-18; First posted 2024-12-24 (Actual); Last update posted 2024-12-24 (Actual); Status verified 2024-12

CONDITIONS: Brain Glioma
MeSH Terms: interventions — Bevacizumab

STUDY DESIGN:
Intervention Model Description: Bevacizumab
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Bevacizumab group (Experimental): Patients were enrolled and given bevacizumab on days 1 and 15, administered by intravenous infusion at 5 mg/kg.
  Interventions: Drug: Bevacizumab

INTERVENTIONS:
Drug: Bevacizumab — Patients were enrolled and given bevacizumab on days 1 and 15, administered by intravenous infusion at 5 mg/kg.

SUMMARY:
Glioblastoma (GBM) usually grows in a diffuse fashion and infiltrates the surrounding brain. The inability to completely excise the tumor often leads to tumor recurrence within a few months of the initial surgery, which ultimately results in the death of the GBM patient.GBM histologically appears to be a tumor of vascular origin characterized by necrosis and microvascular proliferation, and neoangiogenesis is a key factor in the growth and poor prognosis of GBM. Bevacizumab can inhibit the biological effects of VEGF, including the permeability and proliferation of blood vessels, as well as the migration and survival of endothelial cells, so as to inhibit tumor angiogenesis, growth and metastasis. The aim of this study is to evaluate the efficacy and safety of bevacizumab in the preoperative adjuvant treatment of patients with new-onset high-grade gliomas.

DETAILED DESCRIPTION:
Glioblastoma (GBM) usually grows in a diffuse fashion and infiltrates the surrounding brain. The inability to completely excise the tumor often leads to tumor recurrence within a few months of the initial surgery, which ultimately results in the death of the GBM patient.GBM histologically appears to be a tumor of vascular origin characterized by necrosis and microvascular proliferation, and neoangiogenesis is a key factor in the growth and poor prognosis of GBM. Therefore, inhibition of neoangiogenesis has received increasing attention from researchers as an important potential therapeutic target for GBM. Bevacizumab specifically binds to VEGF (mainly to VEGF-A), attenuates or prevents VEGF from binding to VEGFR-1 and VEGFR-2 on the surface of vascular endothelial cells, and blocks VEGFR-mediated downstream signaling pathways, inhibiting their biological activities, reducing tumor neovascularization and limiting tumor growth. Based on this background, the aim of this study was to evaluate the efficacy and safety of bevacizumab in the preoperative adjuvant treatment of patients with new-onset high-grade gliomas.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Male or female.
* Imaging diagnosis of high-grade glioma.
* KPS score ≥60.

Exclusion Criteria:

* Prior treatment with anti-angiogenic targeted drugs;
* Comorbid serious cardiac, pulmonary, hepatic, or renal disease;
* History of an arterial/venous thrombotic event within 6 months prior to screening;
* Combination of infectious diseases such as tuberculosis and viral hepatitis;
* Comorbid infectious diseases such as tuberculosis, viral hepatitis, uncontrolled high blood pressure, bleeding disorders, and long-standing unhealed wounds or incompletely healed fractures;
* Patients with a history of psychotropic substance abuse that cannot be stopped or patients with mental disorders;
* Abnormal coagulation function, with bleeding tendency
* Patients who, in the opinion of the investigator, are not suitable for inclusion in the study (e.g., pregnant and lactating women).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | up to approximately 2 years.
  ORR is defied as the percentage of subject with complete response (CR) or partial response (PR) by investigator assessment per REclsT criteria, version 1.1.

SECONDARY OUTCOMES:
Progression-free survival (PFS) | up to approximately 2 years.
  PFS is defned as the time from randomization untlthe date of first occurence of investigator assessed radiolbgical disease progression or death due to any cause,whichever came first.
Overall survival (OS) | up to approximately 2 years.
  OS is defined as the time from the date of randomization to the date of death due to any cause.
Adverse event (AE) rates | up to approximately 2 years.
  AE assessed by NCI-CTCAE V5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Junkuan Wang, M.D., Principal Investigator — The First Affiliated Hospital of Zhengzhou University
Locations (1):
- The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan, China

IPD SHARING:
Plan to Share IPD: No